CLINICAL TRIAL: NCT02938065
Title: Gastric Emptying of Novel Protein and Carbohydrate Rich Clear Liquids
Brief Title: Gastric Emptying Ultrasound Research Study
Acronym: GERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-0566
Record Dates: First submitted 2016-07-25; First posted 2016-10-19 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Gastric Emptying
MeSH Terms: interventions — High-Energy Shock Waves; Milk

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- 2% Milk (Other): 16 participants will drink 10 ounces of 2% milk Ultrasound scan will be performed at the time of beverage administration and then every 30 minutes thereafter until beverage has been cleared from the stomach
  Interventions: Procedure: Ultrasound; Other: 2% milk
- Apple Juice (Other): 16 participants will drink 10 ounces of apple juice Ultrasound scan will be performed at the time of beverage administration and then every 30 minutes thereafter until beverage has been cleared from the stomach
  Interventions: Procedure: Ultrasound; Other: apple juice
- Ensure Clear (Other): 16 participants will drink 10 ounces of ensure clear Ultrasound scan will be performed at the time of beverage administration and then every 30 minutes thereafter until beverage has been cleared from the stomach
  Interventions: Procedure: Ultrasound; Other: ensure clear

INTERVENTIONS:
Procedure: Ultrasound — Baseline ultrasound is performed upon arrival. Ultrasound is performed when beverage is consumed and then every 30 minutes thereafter until stomach is empty.
Other: 2% milk — 16 participants will drink 10 ounces of 2% milk
  Arms: 2% Milk
Other: apple juice — 16 participants will drink 10 ounces of apple juice
  Arms: Apple Juice
Other: ensure clear — 16 participants will drink 10 ounces of ensure clear
  Arms: Ensure Clear

SUMMARY:
The proposed study will use this technology to observe emptying of the stomach of a protein and carbohydrate rich clear liquid sports/nutrition drink.

DETAILED DESCRIPTION:
In order to ensure safety for elective anesthesia, standard practice requires pre-operative fasting to ensure that the stomach is empty prior to induction. The question of timing of pre-operative consumption of oral fluids remains vexed, and challenges anesthesiologists on a frequent basis. In the past few years, a new controversy in pre-operative fasting has arisen: clear drinks with increased content of protein and carbohydrate have been introduced to the market. Families and professionals alike are confused whether to regard these products as clear liquids (2 hours fasting) or as solids (at least 6 hours).

Ultrasound is now considered an accepted tool in the anesthesia literature as a surrogate for aspiration risk with different materials and in different disease states.

ELIGIBILITY:
Inclusion Criteria:

* 8-14 years old
* Willing to not eat or drink for at least 8 hours overnight beforehand
* Have a BMI < 35

Exclusion Criteria:

* Use tobacco of any kind
* Taking any medications (Females: oral contraceptives okay)
* Suffers from diabetes, Crohn's Disease, Celiac Disease, Malabsorption, Galactosemia
* Has ever has surgery on esophagus, stomach, or small bowel
* Has allergies or intolerances to milk, apple juice, or ensure clear
* Has any surgical condition, disease, or on any medication that could alter stomach emptying rate
* Has any disease that limits day-to-day activities
* Is pregnant or possibly could be pregnant

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Measurement of rate of gastric emptying through measure of the gastric antral cross-sectional area (CSA) | Participants will be followed up to 6 hours after drinking 10 ounces of beverage
Subjective evolution of hunger after ingestion of clear fluids using a validated visual analog scale called the Hunger Satiety Score | Participants will be followed up to 6 hours after drinking 10 ounces of beverage

CONTACTS AND LOCATIONS:
Overall Officials: Jayant Pratap, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Trung Du, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Du T, Hill L, Ding L, Towbin AJ, DeJonckheere M, Bennett P, Hagerman N, Varughese AM, Pratap JN. Gastric emptying for liquids of different compositions in children. Br J Anaesth. 2017 Nov 1;119(5):948-955. doi: 10.1093/bja/aex340. PMID 29077812